CLINICAL TRIAL: NCT06965608
Title: Feasibility Study to Actively Disseminate the Latin America and the Caribbean Code Against Cancer in Primary Healthcare Centers in Aparecida de Goiania (Brazil) - FLACC-Brazil
Brief Title: Feasibility Study to Actively Disseminate the Latin America and the Caribbean Code Against Cancer in Primary Healthcare Centers
Acronym: FLACC-Brazil
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: International Agency for Research on Cancer (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: LACCODE - FLACC-Brazil
Record Dates: First submitted 2025-03-20; First posted 2025-05-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-04

CONDITIONS: Cancer; Latin America and the Caribbean Code Against Cancer (LAC Code)
Keywords: Health Literacy; Cancer Prevention; Health Services Research; Implementation Science; Latin America and the Caribbean Code Against Cancer (LAC Code)
MeSH Terms: conditions — Neoplasms | interventions — Health Personnel

STUDY DESIGN:
Intervention Model Description: Non-randomized four-arm study (before/after pragmatic trial) that will test 2 different implementation strategies either combined or separately for the dissemination of the Latin America and the Caribbean Code Against Cancer within four different primary healthcare units in Aparecida de Goiânia.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Control Group (No Intervention): Participants in this arm will receive no intervention during the study period. They will complete baseline and follow-up assessments to evaluate changes in cancer prevention literacy and health services-related outcomes over time, serving as a comparison for the intervention arms.
- G1: WhatsApp Messaging Intervention - General Population (Experimental): Participants in this arm will receive structured cancer prevention messages via WhatsApp over a four-week period. The messages will cover key recommendations from the Latin America and the Caribbean Code Against Cancer (LAC Code), focusing on actionable steps to reduce cancer risk. Healthcare professionals (HCPs) assigned to this group will not receive any training.
  Interventions: Behavioral: WhatsApp-Based Cancer Prevention Messaging
- G2: Online Workshop for Healthcare Professionals (HCP) (Experimental): Description: Healthcare professionals (HCPs) in this arm will participate in an online, self-paced workshop designed to enhance their knowledge and communication skills related to cancer prevention. The workshop will provide evidence-based training on discussing cancer risk factors and prevention strategies with patients, aligning with the LAC Code recommendations. General population participants assigned to this group will not receive WhatsApp messages.
  Interventions: Behavioral: Online Cancer Prevention Workshop for Healthcare Professionals
- G3: Combined Intervention (WhatsApp + Workshop) (Experimental): This arm will integrate both intervention strategies. General population participants will receive WhatsApp messages with cancer prevention recommendations, while healthcare professionals will complete the online workshop. This combined approach aims to assess whether reinforcing cancer prevention messages at both the community and healthcare provider levels leads to improved outcomes in cancer prevention literacy and health services utilization.
  Interventions: Behavioral: Combined WhatsApp Messaging and Online Workshop

INTERVENTIONS:
Behavioral: WhatsApp-Based Cancer Prevention Messaging — Participants in this group will receive a structured series of WhatsApp messages containing evidence-based cancer prevention recommendations from the Latin America and Caribbean Code Against Cancer (LAC Code). Messages will be delivered over four weeks, 3 times a week, covering key topics such as smoking cessation, healthy diet, physical activity, and regular screening. Engagement metrics will be tracked to assess feasibility and adherence.
  Arms: G1: WhatsApp Messaging Intervention - General Population
Behavioral: Online Cancer Prevention Workshop for Healthcare Professionals — Healthcare professionals assigned to this group will participate in an online workshop designed to improve their knowledge of the LAC Code and communication strategies for cancer prevention counseling. The workshop includes recorded lectures, interactive modules, and knowledge assessments. Completion rates and participant satisfaction will be measured.
  Arms: G2: Online Workshop for Healthcare Professionals (HCP)
Behavioral: Combined WhatsApp Messaging and Online Workshop — Participants in this group will receive both interventions: WhatsApp messages with cancer prevention recommendations and access to the online workshop. The intervention aims to assess whether a combined approach enhances adherence and impact. Engagement with both interventions will be monitored.
  Arms: G3: Combined Intervention (WhatsApp + Workshop)

SUMMARY:
Phase II non-randomized four-arm study (before/after pragmatic trial) that will test 2 different implementation strategies either combined or separately for the dissemination of the Latin America and the Caribbean Code Against Cancer within four different primary healthcare units in Aparecida de Goiânia.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years old)
* Registered at a participating primary healthcare center (UBS) in Aparecida de Goiânia
* Healthcare professionals with at least three months of employment at a participating UBS
* Ability to provide informed consent

Exclusion Criteria:

- Prior diagnosis of any cancer or currently undergoing cancer treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the WhatsApp-Based Intervention | Up to 2 weeks after WhatsApp intervention completion
  Number of participants who report having read at least one WhatsApp message.
Acceptability of the WhatsApp-Based Intervention | Up to 2 weeks after WhatsApp intervention completion
  Mean acceptability score from participant survey (Likert scale 1-5) evaluating message usefulness and clarity.
Appropriateness of the WhatsApp-Based Intervention | Up to 2 weeks after WhatsApp intervention completion
  Proportion of participants who indicate willingness to receive similar messages in the future (Yes/No).

OTHER OUTCOMES:
Receipt of Cancer Prevention Counseling Among the General Population (KAS Questionnaire) | Baseline and final assessment (up to 2 weeks after intervention)
  Proportion of general population participants reporting receipt of at least one type of cancer prevention counseling (e.g., smoking cessation, diet, physical activity) as assessed by the KAS questionnaire
Intention to Provide Cancer Prevention Counseling Among Healthcare Professionals (KAP Questionnaire) | Baseline, post-workshop (up to 2 weeks), and final assessment (up to 2 weeks after intervention)
  Proportion of healthcare professionals reporting intention to integrate cancer prevention counseling into clinical practice, assessed via the KAP questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- HMAP - Hospital Municipal de Aparecida de Goiânia, Aparecida de Goiânia, Goiás, Brazil

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to privacy considerations and institutional policies governing data access. However, aggregated and de-identified study results will be shared through peer-reviewed publications and conference presentations.

REFERENCES:
- [Background] Busetto L, Wick W, Gumbinger C. How to use and assess qualitative research methods. Neurol Res Pract. 2020 May 27;2:14. doi: 10.1186/s42466-020-00059-z. eCollection 2020. PMID 33324920
- [Background] Espina C, Feliu A, Gonzalez Vingut A, Liddle T, Jimenez-Garcia C, Olaya-Caro I, Perula-De-Torres LA. Population-Based Cancer Prevention Education Intervention Through mHealth: A Randomized Controlled Trial. J Med Syst. 2024 Jan 9;48(1):9. doi: 10.1007/s10916-023-02026-y. PMID 38194118
- [Background] Delucchi KL, Tajima B, Guydish J. Development of the Smoking Knowledge, Attitudes, and Practices (S-KAP) Instrument. J Drug Issues. 2009 Mar;39(2):347-364. doi: 10.1177/002204260903900207. PMID 20717496
- [Background] Nardi A, Mitrova S, Angelici L, De Gregorio CG, Biliotti D, De Vito C, Vecchi S, Davoli M, Agabiti N, Acampora A. Developing a Questionnaire Evaluating Knowledge, Attitudes and Behaviors on Audit & Feedback among General Practitioners: A Mixed Methods Study. Healthcare (Basel). 2023 Apr 24;11(9):1211. doi: 10.3390/healthcare11091211. PMID 37174753
- [Background] Patsopoulos NA. A pragmatic view on pragmatic trials. Dialogues Clin Neurosci. 2011;13(2):217-24. doi: 10.31887/DCNS.2011.13.2/npatsopoulos. PMID 21842619
- [Background] Espina C, Feliu A, Maza M, Almonte M, Ferreccio C, Finck C, Herrero R, Dommarco JR, de Almeida LM, Arrossi S, Garcia PJ, Garmendia ML, Mohar A, Murillo R, Santamaria J, Tortolero-Luna G, Cazap E, Gabriel OO, Paonessa D, Zoss JW, Luciani S, Carvalho A, Schuz J; Working Groups of Scientific Experts. Latin America and the Caribbean Code Against Cancer 1st Edition: 17 cancer prevention recommendations to the public and to policy-makers (World Code Against Cancer Framework). Cancer Epidemiol. 2023 Oct;86 Suppl 1:102402. doi: 10.1016/j.canep.2023.102402. Epub 2023 Oct 16. PMID 37852725
- [Background] Fleary SA, Paasche-Orlow MK, Joseph P, Freund KM. The Relationship Between Health Literacy, Cancer Prevention Beliefs, and Cancer Prevention Behaviors. J Cancer Educ. 2019 Oct;34(5):958-965. doi: 10.1007/s13187-018-1400-2. PMID 30022378
- [Background] Morris NS, Field TS, Wagner JL, Cutrona SL, Roblin DW, Gaglio B, Williams AE, Han PJ, Costanza ME, Mazor KM. The association between health literacy and cancer-related attitudes, behaviors, and knowledge. J Health Commun. 2013;18 Suppl 1(Suppl 1):223-41. doi: 10.1080/10810730.2013.825667. PMID 24093358
- [Background] Strasser-Weippl K, Chavarri-Guerra Y, Villarreal-Garza C, Bychkovsky BL, Debiasi M, Liedke PE, Soto-Perez-de-Celis E, Dizon D, Cazap E, de Lima Lopes G Jr, Touya D, Nunes JS, St Louis J, Vail C, Bukowski A, Ramos-Elias P, Unger-Saldana K, Brandao DF, Ferreyra ME, Luciani S, Nogueira-Rodrigues A, de Carvalho Calabrich AF, Del Carmen MG, Rauh-Hain JA, Schmeler K, Sala R, Goss PE. Progress and remaining challenges for cancer control in Latin America and the Caribbean. Lancet Oncol. 2015 Oct;16(14):1405-38. doi: 10.1016/S1470-2045(15)00218-1. PMID 26522157
- [Background] Barrios CH, Werutsky G, Mohar A, Ferrigno AS, Muller BG, Bychkovsky BL, Castro E CJ, Uribe CJ, Villarreal-Garza C, Soto-Perez-de-Celis E, Gutierrez-Delgado F, Kim JS, Ismael J, Delgado L, Santini LA, Teich N, Chavez PC, Liedke PER, Exman P, Barroso-Sousa R, Stefani SD, Caceres SAB, Rebelatto TF, Pastrana T, Chavarri-Guerra Y, Vargas Y, Cazap E. Cancer control in Latin America and the Caribbean: recent advances and opportunities to move forward. Lancet Oncol. 2021 Nov;22(11):e474-e487. doi: 10.1016/S1470-2045(21)00492-7. PMID 34735817
- [Background] Rezende LFM, Lee DH, Louzada MLDC, Song M, Giovannucci E, Eluf-Neto J. Proportion of cancer cases and deaths attributable to lifestyle risk factors in Brazil. Cancer Epidemiol. 2019 Apr;59:148-157. doi: 10.1016/j.canep.2019.01.021. Epub 2019 Feb 14. PMID 30772701
- See also: GLOBOCAN — https://gco.iarc.who.int/today